CLINICAL TRIAL: NCT03838835
Title: Equine Facilitated Cognitive Behavioral Therapy (CBT) Group Therapy for Youth Anxiety
Brief Title: Equine Facilitated CBT Group Therapy for Youth Anxiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01424
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Equine-facilitated group therapy (Experimental)
  Interventions: Behavioral: TAU is equine-facilitated group therapy
- Augmented equine-facilitated CBT group program (Experimental)
  Interventions: Behavioral: Augmented equine-facilitated CBT group program
- Wait List Control (WLC) (Other)
  Interventions: Other: WLC

INTERVENTIONS:
Behavioral: Augmented equine-facilitated CBT group program — Consists of CBT strategies including 1) providing psychoeducation about anxiety, 2) teaching coping strategies when anxious,and 3) identifying and addressing dysfunctional thoughts that maintain anxiety.
  Arms: Augmented equine-facilitated CBT group program
Behavioral: TAU is equine-facilitated group therapy — TAU is equine-facilitated group therapy at GallopNYC, which consists of horseback riding and integrates strategies to support the development of cognitive, physical, emotional, and social skills.
  Arms: Equine-facilitated group therapy
Other: WLC — WLC consists of youth who are not yet receiving any services at Gallop NYC.
  Arms: Wait List Control (WLC)

SUMMARY:
The purpose of this study is to evaluate a 10-week equine facilitated cognitive behavioral therapy (CBT) group program for youth between ages of 6 to 17 with symptoms of anxiety. The program will be delivered at GallopNYC, a stable that provides equine-facilitated group therapy to youth with a range of mental health problems.

DETAILED DESCRIPTION:
The equine-facilitated group therapy normally provided at GallopNYC (Treatment as Usual, TAU) will be compared to an augmented group program that will include CBT strategies, including psychoeducation to the child and caregiver about anxiety, coping strategies to use when anxious, and identifying and addressing dysfunctional thoughts that maintain anxiety. Seventy-five children between 6 to 17 years of age will be randomized to TAU (equine-facilitated group therapy), the augmented group therapy that contains CBT strategies, or wait list control. Outcomes include anxiety symptoms, self-efficacy,receipt of services, functioning and the child's relationship with the horse.

ELIGIBILITY:
Inclusion Criteria:

* A child aged 6-17 seeking services for anxiety at Gallop NYC, who (based on the screener administered by GallopNYC) evidence symptoms of anxiety (as measured by a score of 2 or more on the GAD 2 item questionnaire) and a minimum functioning score of 51 (as measured by the child global assessment scale)
* Caregivers will also serve as study respondents. To do so, they must meet the following criteria:
* Primary caregiver/ legal guardian of a child who meets eligibility criteria
* Aged 18 years or older
* English speaking

Providers will serve as study therapists. To do so, they must meet the following criteria:

* PATH-certified provider employed at Gallop NYC

Exclusion Criteria:

* Inability to provide informed consent
* Child does not meet criteria for anxiety symptoms (as measured by a score of 2 or more on the GAD 2 item questionnaire) and/or does not meet minimum level of functioning (does not meet a minimum functioning score of 51 as measured by the child global assessment scale)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Anxiety, as measured by the SCARED | Baseline to 10 Weeks
  41 item questionnaire scored on a 3-point Likert Scale ranging from "not true" to "very true." Items are summed, with higher scores indicating more anxiety symptoms (a cutoff of 25 indicates an anxiety disorder).

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Hoagwood, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States